CLINICAL TRIAL: NCT03012464
Title: Pathologic and Functional Assessment of Rectal Prolapse in Young Patients
Brief Title: Pathologic Assessment of Rectal Prolapse in the Young
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Other Study IDs: mansourau2017
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pathologic and functional assessment: Patients of both genders, aging below 45 years with internal or external rectal prolapse
  Interventions: Other: Pathologic and functional assessment

INTERVENTIONS:
Other: Pathologic and functional assessment — Random biopsies will be taken from the pelvic floor muscles, external anal sphincter, and the lateral supportive ligaments of the rectum during surgical treatment of rectal prolapse whether via the abdominal or perineal approach. Tissue samples will be subjected to immunohistochemistry to calculate the ratio between collagen type I and type III, and to reveal any myopathic or degenerative changes

SUMMARY:
Patients aging less than 45 years with rectal prolapse will undergo full pathologic and functional assessment to determine the underlying etiology.

DETAILED DESCRIPTION:
Full clinical assessment of the patients will be conducted by history taking querying the type and duration of symptoms, associated medical conditions, history of previous surgery for rectal prolapse, and presence of fecal incontinence which will be graded by Wexner continence score. In addition, patients will undergo thorough general and local examination to determine the type of rectal prolapse (internal or external) and the condition of the anal sphincters and pelvic floor muscles.

Functional assessment of the anorectal region will be done by anal manometry to measure the resting and squeeze anal pressures, rectal sensation and compliance; endorectal ultrasonography to assess the integrity of the anal sphincters; and pudendal nerve terminal motor latency (PNTML) to exclude pudendal neuropathy.

Random biopsies (2-4 in number) will be taken from the pelvic floor muscles, external anal sphincter, and the lateral supportive ligaments of the rectum during surgical treatment of rectal prolapse whether via the abdominal or perineal approach. Tissue samples will be preserved in formalin solution and will be sent for histopathological examination. Tissue samples will be subjected to immunohistochemistry to calculate the ratio between collagen type I and type III, and to reveal any myopathic or degenerative changes. Additionally, schistosomal affection of the pelvic floor muscles will be detected by immunohistochemistry examination for the ova of schistosomal mansoni.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aging below 45 years with primary or recurrent rectal prolapse, whether internal or external prolapse

Exclusion Criteria:

* Patients above 45 years, patients with associated anorectal pathology as anal fissure, hemorrhoids or neoplasm, and patients with documented psychiatric or mental disorders.

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients of both genders aging below 45 years with primary or recurrent rectal prolapse, whether internal or external prolapse, will be included. Patients above 45 years, patients with associated anorectal pathology as anal fissure, hemorrhoids or neoplasm, and patients with documented psychiatric or mental disorders will be excluded
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Collagen I:III ratio | immediate after surgery
  Pathologic assessment of the taken biopsies to examine the ratio between collagen type I and type III

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University
Locations (2):
- Egypt (2):
  - Mansoura University hospitals, Al Mansurah, Dakahlia Governorate
  - Mansoura university hospital, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD